CLINICAL TRIAL: NCT03093168
Title: A Phase I Clinical Trial of T-Cells Targeting B-Cell Maturation Antigen for Subjects With BCMA-positive Multiple Myeloma
Brief Title: BCMA Chimeric Antigen Receptor Expressing T Cells in Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other)
Collaborators: Hrain Biotechnology Co., Ltd. (Industry); First Affiliated Hospital of Wenzhou Medical University (Other); Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: anti-BCMA CART
Record Dates: First submitted 2017-03-15; First posted 2017-03-28 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-BCMA CAR-T (Experimental): Administration of anti-BCMA:TCRζ-4-1-BB CAR-T cells to patients with multiple myeloma
  Interventions: Biological: Anti-BCMA CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Anti-BCMA CAR-T cells — Retroviral vector-transduced autologous T cells to express anti-BCMA CAR
Drug: Fludarabine — dose: 25mg/m2/d
Drug: Cyclophosphamide — Dose: 40mg/kg

SUMMARY:
The goal of this clinical trial is to study the feasibility and efficacy of anti-B-Cell Maturation Antigen (BCMA) expressing T cells in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine the feasibility ad safety of BCMA CAR-T cells in treating patients with multiple myeloma.
2. To determine in vivo dynamics and persistency of BCMA CAR-T cells.
3. To access the efficacy of BCMA CAR-T cells in patients with multiple myeloma.

Secondary Objectives

1. To assess the bone marrow and tumor migration of BCMA CAR-T cells.
2. To investigate the tumor killing capability of BCMA CAR-T cells in vitro
3. To investigate the possibility of host immune response to the mouse derived BCMA scFv, and evaluate its correlation to CAR-T persistence.
4. To correlate the subsets and differentiation of BCMA CAR-T cells to observed anti-tumor efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Expected survival > 12 weeks
* Diagnosis of Multiple Myeloma by MWG criteria 20
* Patients previously received at least 3 different prior treatment regimens for multiple myeloma, including alkylating agent, protein inhibitors, and immunomodulator, and have disease progression in the past 60 days
* Important organs function enough to tolerate this therapy
* At least 90 days after stem cell transplantation
* Clinical performance status of ECOG score 0-4
* Accessible to intravenous injection, and no white blood cell collection contraindications
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 30 days after the CTL infusion. Male partner should use a condom
* Able to understand and sign the Informed Consent Document.

Exclusion Criteria:

* Patients with symptoms of central nervous system
* Patients with second malignancies in addition to multiple myeloma
* Active hepatitis B or C, HIV infections
* Any other active diseases could affect the enrollment of this trial
* Suffering severe cardiovascular or respiratory disease
* Poorly controlled hypertension
* Long term use of immunosuppressive agents after organ transplantation, except currently receiving or recently received glucocorticoid treatment
* A history of mental illness and poorly controlled
* Screening showing target cell transduction efficacy is lower than 30%, or T cell proliferation is not enough for infusion (less than 5 fold)
* Occurrence of unstable pulmonary embolism, deep vein thrombosis, or other major arterial/venous thromboembolic events 30 days prior to assignment
* Women of child-bearing potential who are pregnant or breastfeeding during therapy, or have a planned pregnancy with 2 months after therapy
* Women of child-bearing potential who are not willing to practice birth control from the time of enrollment on this study and for 2 months after receiving the preparative regimen. Women of child bearing potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
* Active systemic infections or uncontrolled infection within 14 days prior enrollment
* Subjects suffering disease affects the understanding of informed consent or complying with study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0 | 6 months
  Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0

SECONDARY OUTCOMES:
Overall complete remission rate defined by the standard response criteria for malignant lymphoma for each arm | 8 weeks
  Overall complete remission rate defined by the standard response criteria for malignant lymphoma for each arm
Duration of CAR-positive T cells in circulation | 6 months
  Duration of CAR-positive T cells in circulation
Total number of CAR-positive T cells infiltrated into lymphoma tissue | 6 months
  Total number of CAR-positive T cells infiltrated into lymphoma tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Province of TCM, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zhou L, Fu W, Wu S, Xu K, Qiu L, Xu Y, Yan X, Zhang Q, Zhang M, Wang L, Hong R, Chang AH, Yu J, Fu S, Kong D, Li L, Wang Y, Li Z, Jiang H, Huang J, Liu Z, Su N, Wei G, Hu Y, Huang H. Derivation and validation of a novel score for early prediction of severe CRS after CAR-T therapy in haematological malignancy patients: A multi-centre study. Br J Haematol. 2023 Aug;202(3):517-524. doi: 10.1111/bjh.18873. Epub 2023 May 16. PMID 37192741